CLINICAL TRIAL: NCT01151917
Title: Identification of a Novel Factor(s) of Importance to Insulin Resistance -Repeated Blood Sampling Before and After Biliopancreatic Diversion
Brief Title: Proteomics in Morbid Obesity After Bariatric Surgery
Acronym: PROTOBESE
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, professor, Catholic University of the Sacred Heart
Other Study IDs: UCSC
Record Dates: First submitted 2010-06-11; First posted 2010-06-29 (Estimated); Last update posted 2014-01-30 (Estimated); Status verified 2014-01

CONDITIONS: Insulin Resistance; Proteomics; Morbid Obesity
Keywords: Bilio-pancreatic diversion; morbid obesity; insulin resistance; proteomics
MeSH Terms: conditions — Insulin Resistance; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma samples at fasting and after a meal
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bilio-pancreatic diversion: Each subject is own control

SUMMARY:
Glycemic control is rapidly restored in patients with insulin resistance after bariatric surgery, in particular after the mal-absorptive one (i.e. Bilio-pancreatic diversion, BPD). To evaluate the mechanisms allowing restoration of insulin sensitivity after BPD the investigators aimed at identifying by using a proteomic approach plasma proteins or peptides that may be involved in the remarkably fast and explicit restoration of insulin sensitivity. In addition to the unbiased proteomics approach, a selection of recognized markers for metabolic control will be measured. These efforts all aim at an increased understanding of how insulin sensitivity is regulated and may provide novel ideas of how to treat insulin resistance and type 2-diabetes.

DETAILED DESCRIPTION:
Study design The study is designed as a single-centre, observational study. The patients will undergo routine analyses usually performed before and after biliopancreatic diversion surgery (BPD), independently of the participation to this specific protocol with the only exception of meal test. Twenty morbidly obese male subjects scheduled for BPD for will be included in the study.

The inclusion and exclusion criteria are set as to create a sufficiently homogenous study population.

As outlined in the study flow chart subjects will be studied and blood samples collected at 3 weeks (+/- 1 week) and 4 days (+/- 1 day) before the day of BPD surgery (baseline-1 and baseline-2), at the day of surgery (day 0), every second day after surgery during the first week (immediate post surgery) as well as two and four weeks after surgery (post surgery-1 and post surgery-2). A deviation of +/- 2 days is allowed for the post surgery-1 and post surgery-2 visits.

All fasting samples are obtained in the morning after an overnight fast (12 h). Immediate post surgery (fasting) samples will be collected after 12 h rest from parenteral nutrition from the arm not used for nutritional substitution during the first 4 days after surgery (when parenteral nutrition is given). The immediate post surgery (fasting) samples obtained from day 5 and forward after surgery, when subjects have started to eat, will be obtained in the morning after an overnight fast (12 h). Nutrient stimulation samples will be obtained at baseline-1 and 2 and post surgery-1 and 2 after intake of a test meal. A complete list of all procedures for each visit is provided in Table 1 and an overview of all planned blood samples, including volumes and purpose is provided in Table 2. Motivations for the collection of various samples are provided under section 10.3.1 "Proteomics analysis, experimental design issues".

In case of discontinuation, additional subjects should be enrolled such that a complete set of samples from no less than 20 subjects can be obtained.

Target subject population Inclusion criteria

* Morbidly obese male with a BMI >40 kg/m2 who, for their obesity disease, are eligible for bariatric surgery and have accepted to undergo BPD
* Confirmed insulin resistance; fasting serum insulin level > 60 pmol/L
* Age 25-55 years
* Weight stable for at least 6 months before the study (+/- 5 kg within the previous 6 months)
* Stable medication
* Provision of informed consent, statistical analysis, and publications of obtained results Exclusion criteria
* Patients not eligible for BPD
* Incapacity to give a valid informed consent or unwilling to give the consent
* Patients eligible for BPD, but with:

  * Type 2-diabetes mellitus
  * Significant illness within the two weeks preceding surgery, as judged by the physician.
  * Obvious infection (bacteria, virus etc)
  * Major cardiovascular disease
  * Major gastrointestinal, respiratory, or any hormonal disorders
  * Medication affecting lipid metabolism within 3 months of the study
  * History of drug addiction and/or alcohol use
  * Suspected or confirmed poor compliance
  * Exercise +/-3 times a week
  * Blood donation within 12 weeks preceding screening visit

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese male with a BMI >40 kg/m2 who, for their obesity disease, are eligible for bariatric surgery and have accepted to undergo BPD
* Confirmed insulin resistance; fasting serum insulin level > 60 pmol/L
* Age 25-55 years
* Weight stable for at least 6 months before the study (+/- 5 kg within the previous 6 months)
* Stable medication
* Provision of informed consent, statistical analysis, and publications of obtained results

Exclusion Criteria:

* Patients not eligible for BPD
* Incapacity to give a valid informed consent or unwilling to give the consent
* Patients eligible for BPD, but with:

  * Type 2-diabetes mellitus
  * Significant illness within the two weeks preceding surgery, as judged by the physician.
  * Obvious infection (bacteria, virus etc)
  * Major cardiovascular disease
  * Major gastrointestinal, respiratory, or any hormonal disorders
  * Medication affecting lipid metabolism within 3 months of the study
  * History of drug addiction and/or alcohol use
  * Suspected or confirmed poor compliance
  * Exercise +/-3 times a week
  * Blood donation within 12 weeks preceding screening visit

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Twenty male, morbidly obese subjects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Proteomics | 2 years
  used to identify plasma proteins or peptides that may be involved in the remarkably fast and explicit restoration of insulin sensitivity seen in morbidly obese patients with insulin resistance shortly after gastric bypass surgery by BPD.

SECONDARY OUTCOMES:
Insulin sensitivity and secretion and incretins | 2 years
  Selection of recognized markers for metabolic control. Insulin secretion is measured by C-peptide deconvolution and insulin sensitivity by minimal modelling of glucose-insulin after a meal. Increatins will be measured too.

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, Professor, Principal Investigator — Catholic University of Rome
Locations (1):
- Day Hospital of Metabolic Diseases, Catholic University, Rome, Italy

REFERENCES:
- [Derived] Karlsson C, Wallenius K, Walentinsson A, Greasley PJ, Miliotis T, Hammar M, Iaconelli A, Tapani S, Raffaelli M, Mingrone G, Carlsson B. Identification of Proteins Associated with the Early Restoration of Insulin Sensitivity After Biliopancreatic Diversion. J Clin Endocrinol Metab. 2020 Nov 1;105(11):e4157-68. doi: 10.1210/clinem/dgaa558. PMID 32830851